CLINICAL TRIAL: NCT04529486
Title: Effects of Kinesio Taping on Upper Extremity Functionality in Participants With Cerebral Palsy
Brief Title: Kinesio Taping in Cerebral Palsy Upper Extremity Functionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, Associated Proffesor, Baskent University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KA20/46
Record Dates: First submitted 2020-08-21; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Cerebral Palsy
Keywords: Kinesiotape; Cerebral palsy; upper extremity functionality
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The children with Cerebral Palsy included in this study consisted of 2 groups, the study group and the control group. No application was made to the control group. The same participant group was included as the experimental group after 1 week of rest. The assessments were done three times for each group (beginning - 45min later - 1 week later)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Kinesio taping (Experimental): Kinesio taping was applied to the study group to improve posture and improve function in the shoulder area. Measurements were carried out for the study group before and after application (with tape on). The tape was then removed and the measurements were repeated after 1 week.
  Interventions: Other: Kinesio taping
- Group 2: Control (No Intervention): No application was made to the control group.

INTERVENTIONS:
Other: Kinesio taping — Before applying the tape, it was checked whether the children were allergic. Tape was first started from the distal part of the fingers and taped with 0% tension with Kinesio Taping Functional Correction Technique. Another I tape was applied from palmar area of the hand to spina scapula for supination of the forearm and external rotation of the shoulder with %0 tension to make functional correction (Figure 2). Kinesio Taping Functional Correction method is suggested to be done with 75% of tension but for children, we applied it with 0% tension to minimize the shear effects to the skin4. Kinesio Tex Light Touch Plus tape was used for taping application (Kinesio Co., USA).
  Arms: Group 1: Kinesio taping

SUMMARY:
Purpose: The aim of this study is to investigate the effects of kinesio taping on upper extremity functionality in participants with Cerebral Palsy.

Methods: This study included 14 children aged 6-16 years, diagnosed with Cerebral Palsy. The children with Cerebral Palsy were divided into 2 groups, the study group and the control group. Assessments were done three times for each group (beginning - 45min later - 1 week later). Frenchay Arm Test was used to evaluate upper extremity functionality in participants with Cerebral Palsy. Kinesio taping was applied to study group to improve posture and function in shoulder area.

ELIGIBILITY:
Inclusion criteria were as follows;

* To have a cognitive level to comprehend the instructions
* Not having a cooperative problem that may prevent communication
* Continuing special education regularly Exclusion criteria were as follows;
* Those with orthopedic problems
* Any surgical procedure
* Participants with cognitive problems
* Participants who do not regularly receive physiotherapy

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Upper extremity functionality | 2 weeks
  Frenchay Arm Test was used to evaluate upper extremity functionality in participants with Cerebral Palsy.
  Frenchay Arm Test: The total duration of the test is 3 minutes. Each task is scored as 1 point. The participant takes minimum 0 and maximum 5 points. Higher scores indicate better functionality. The participant sits in the chair with a table in front of him and puts his hands on his knees and tries to perform the following sequential tasks with the affected arm / hand.
  1. Fixing the ruler 2. Holding a roller 3. Raising the cup 4. Attaching a latch to the bar 5. Combing hair

CONTACTS AND LOCATIONS:
Overall Officials: Nihan O Pekyavas, Principal Investigator — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No